CLINICAL TRIAL: NCT00708591
Title: A Phase Ib Study Administering Rapamycin (Sirolimus) With Ketoconazole in Patients With Advanced Malignancies
Brief Title: Study of Rapamycin Plus Ketoconazole in Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13274B
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Sirolimus; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Rapamycin; Drug: Ketoconazole

INTERVENTIONS:
Drug: Rapamycin — Oral Rapamycin once weekly at assigned dose in 4 week cycles. Dosing can continue until disease progression or severe side effects are seen.
  Other Names: Rapamune; Sirolimus
Drug: Ketoconazole — Twice daily (200mg each time) at the start of the second week of therapy for 4 consecutive days. Dosing continues every week after the second week of therapy.

SUMMARY:
To determine the maximum tolerated dose, observed toxicities, and dose limiting toxicities, and antitumor response of rapamycin plus ketoconazole in patients with advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Patients with hematologic malignancies (lymphoma, multiple myeloma and CLL only) are eligible to participate in the phase Ib portion of the trial only
* At least 4 weeks since prior chemotherapy or radiation therapy (6 weeks if the last regimen included BCNU or mitomycin C).
* Age >18 years.
* ECOG performance status less than or equal to 2
* Life expectancy of more than 3 months.
* Normal organ and marrow function as defined below:

  * Hemoglobin ≥ 10 g/dl
  * Leukocytes ≥ 3,000/µL

    o WBC ≥ 1,500/µL for patients with hematologic malignancies
  * Absolute neutrophil count ≥ 1,500/µL (≥ 1,000/µL for patients with hematologic malignancies)
  * Absolute lymphocyte count ≥1000/µL
  * Platelets ≥ 100,000/µL (≥ 50,000/µL for patients with hematologic malignancies)
  * Total bilirubin within normal institutional limits
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 times institutional ULN
  * Serum triglycerides ≤ 500 mg/dl
  * Creatinine within normal institutional limits OR
  * Creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Able to understand and the willing to sign a written informed consent document.

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Receiving any other investigational agents.
* Uncontrolled brain metastases or malignancy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to rapamycin.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Severe immunodeficient state (as judged by the treating physician)
* Pregnancy (breast-feeding must be discontinued)
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with rapamycin.
* Concurrent use of cyclosporine, tacrolimus, and rifampin, terfenadine, astemizole, cisapride, rosiglitazone or pioglitazone due to possible interactions with the study drugs. Ketoconazole cannot be taken within 2 hours of an antacid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 4 weeks

SECONDARY OUTCOMES:
observed toxicities | 4 weeks
anti-tumor response | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States